CLINICAL TRIAL: NCT04526223
Title: Allogeneic HCT Outcomes in MF Patients Exposure to Ruxolitinib During Transplantation
Brief Title: Outcomes of MF Patients Exposure to Ruxolitinib During Transplantation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: xuna (Other)
Responsible Party: Sponsor-Investigator, xuna, doctor, Nanfang Hospital, Southern Medical University
Organization: Nanfang Hospital, Southern Medical University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HSCT-MF-01
Record Dates: First submitted 2020-02-16; First posted 2020-08-25 (Actual); Last update posted 2022-04-15 (Actual); Status verified 2022-04

CONDITIONS: Time of Hematopoietic Reconstruction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- treatment group (Experimental): MF patients exposure to ruxolitinib during transplantation
  Interventions: Other: comprehensive treatment regimen

INTERVENTIONS:
Other: comprehensive treatment regimen — 1. Diagnosis MF(includ Post-ET,Post-PV,PMF，MDS/MPN with MF)
  2. With at least two month Ruxolitinib treatment prior to transplantation
  3. DAC+BF as myeloablative conditioning regimen
  4. received Rux at +5d in ASCT and continued to +60d

SUMMARY:
Increasing experience of Ruxolitinib pre-allo SCT and data concerning Ruxolitinib during transplantation

1. Diagnosis MF(includ Post-ET,Post-PV,PMF,MDS/MPN with MF)
2. With at least two month Ruxolitinib treatment prior to transplantation
3. DAC+BF as myeloablative conditioning regimen
4. CSA from day -3 and MMF from day +1 until day 28 ATG Neovii® at dose of 7.5mg/KG for mismatch donor
5. received Rux at +6d in ASCT and continued to +60d

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-60 years old, gender is not limited;
2. Diagnosis MF(includ Post-ET,Post-PV,PMF) according to 2016 WHO
3. With at least two month Ruxolitinib treatment before transplantation
4. Informed consent of the patient or his legal representative

Exclusion Criteria:

1. HCT-CI score≥2
2. Woman who is pregnant or nursing
3. MPN Patients who have received allogeneic hematopoietic stem cell transplantation

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2017-04-20 (Actual); Primary Completion 2022-12-20 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Time of neutrophils reconstruction | 1 year
  Neutrophils count≧0.5G/L without G-CSF

SECONDARY OUTCOMES:
The incidence rate of GVHD | 1 year
  The incidence rate of aGVHD and cGVHD

CONTACTS AND LOCATIONS:
Overall Officials: H Nanfang, doctor, Principal Investigator — Nanfang Hospital, Southern Medical University
Locations (1):
- NanfangH, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Barbui T, Tefferi A, Vannucchi AM, Passamonti F, Silver RT, Hoffman R, Verstovsek S, Mesa R, Kiladjian JJ, Hehlmann R, Reiter A, Cervantes F, Harrison C, Mc Mullin MF, Hasselbalch HC, Koschmieder S, Marchetti M, Bacigalupo A, Finazzi G, Kroeger N, Griesshammer M, Birgegard G, Barosi G. Philadelphia chromosome-negative classical myeloproliferative neoplasms: revised management recommendations from European LeukemiaNet. Leukemia. 2018 May;32(5):1057-1069. doi: 10.1038/s41375-018-0077-1. Epub 2018 Feb 27. PMID 29515238
- [Background] Kroger N, Shahnaz Syed Abd Kadir S, Zabelina T, Badbaran A, Christopeit M, Ayuk F, Wolschke C. Peritransplantation Ruxolitinib Prevents Acute Graft-versus-Host Disease in Patients with Myelofibrosis Undergoing Allogenic Stem Cell Transplantation. Biol Blood Marrow Transplant. 2018 Oct;24(10):2152-2156. doi: 10.1016/j.bbmt.2018.05.023. Epub 2018 May 22. PMID 29800615
- [Background] Shahnaz Syed Abd Kadir S, Christopeit M, Wulf G, Wagner E, Bornhauser M, Schroeder T, Crysandt M, Mayer K, Jonas J, Stelljes M, Badbaran A, Ayuketang Ayuk F, Triviai I, Wolf D, Wolschke C, Kroger N. Impact of ruxolitinib pretreatment on outcomes after allogeneic stem cell transplantation in patients with myelofibrosis. Eur J Haematol. 2018 Sep;101(3):305-317. doi: 10.1111/ejh.13099. Epub 2018 Jul 4. PMID 29791053
- [Background] Jagasia M, Zeiser R, Arbushites M, Delaite P, Gadbaw B, Bubnoff NV. Ruxolitinib for the treatment of patients with steroid-refractory GVHD: an introduction to the REACH trials. Immunotherapy. 2018 Apr;10(5):391-402. doi: 10.2217/imt-2017-0156. Epub 2018 Jan 10. PMID 29316837